CLINICAL TRIAL: NCT05230953
Title: Fourth COVID-19 Vaccine Dose- mRNA1273 - the Sheba HCW Cohort
Brief Title: Fourth COVID-19 Vaccine Dose- mRNA1273
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Gili Regev-Yochay MD, Director of Infection Prevention & Control Unit, Sheba Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9035-21
Record Dates: First submitted 2022-02-02; First posted 2022-02-09 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: COVID-19 Pandemic
Keywords: COVID-19; mRNA1273; Omicron; immunogenicity
MeSH Terms: conditions — COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Intervention Model Description: This is a prospective intervention study, to test the effect of a 4th dose, by comparing the immune response before and after the 4th dose, given to 150-200 volunteers, as well as comparing their responses with (1) a control group of individuals vaccinated with 3 doses but without the 4th. (2) a similar group vaccinated with BNT162b2 as a 4th dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 4th dose mRNA1273 vaccine (Experimental): The investigators will recruit 150-200 volunteers, who received the 3rd dose at least 4 months previously, and have a known serology history (showing an immune response (even if just a low response) to the three previous doses, but with a recent relatively low IgG (below 700 BAU). These volunteers will recieve a 4th dose (50microgram) of the mRNA1273 vaccine
  Interventions: Biological: mRNA1273 vaccine
- Control (No Intervention): As controls, a sub-cohort of similar HCW, who are recruited to the Sheba COVID Cohort study (IRB 8008-20) and are followed monthly with serology tests, and are not receiving the 4th dose. The control group, all of whom signed an informed consent and allowed blood samples to be used for further immunologic studies, will be matched by age, gender, time from 3rd vaccine dose and IgG titers, and will be followed similarly
- 4th dose BNT162b2 vaccine (Experimental): The outcomes will be compared to those participating in study IRB-8980-21, with a similar protocol, initiated 1 week earlier.
  Interventions: Biological: mRNA1273 vaccine

INTERVENTIONS:
Biological: mRNA1273 vaccine — fourth dose of the mRNA1273 vaccine (50 microgram) adminstered IM
  Arms: 4th dose BNT162b2 vaccine; 4th dose mRNA1273 vaccine

SUMMARY:
The Omicron variant of concern (VOC) is currently rapidly spreading worldwide, with extremely high transmission rates, with an estimated R of >3.

The investigators now have preliminary, yet unpublished data, showing slow waning of the immune response after the third dose of the BNT162b2 mRNA vaccine within 4 months after this dose . While these data would not have been worrisome in the Delta VOC era, this may be different with the emergence of the Omicron VOC.

These data raise the question of when and will a 4th dose be needed to cope with the emergence of Omicron. However, if a maximal effect of the current vaccine has been reached against Omicron, with a third dose, will a 4th dose have any added value? Here, the investogators will study the potential immunogenicity of a 4th dose, together with assessing safety and effectiveness in preventing infections

DETAILED DESCRIPTION:
The aim of the study is to assess the immunogenicity of a 4th dose, and its durability. This will be measured by following IgG, IgA, Pseudoneutralization assays, microneutralization, avidity, T-cell activity and B-cell repertoire and comparing them to a matched control group, who are participating in the Sheba COVID Cohort study. The investigators will also assess safety and vaccine effectiveness by active surveillance of adverse events and by following incidence of SARS-CoV-2 infections.

This is a prospective intervention study, to test the effect of a 4th dose of a heterologeous vaccine (mRNA1273, following 3 doses of BNT162b2), by comparing the immune response before and after the 4th dose, given to 150-200 volunteers, as well as comparing their responses with a (1) control group of individuals vaccinated with 3 doses but without the 4th (2) an arm of similar study with a 4th dose of BNT162b2 (homologeous vaccine). All study participants would be health care workers from Sheba medical Center, who are participating in the Sheba COVID Cohort study and have a serology test from the previous 3 months. Participation in the study will be confidential and will not be disclosed to the worker's direct supervisor. For this study, the investigators will recruit 150-200 volunteers, who received the 3rd dose at least 4 months previously, and have a known serology history (showing an immune response (even if just a low response) to the three previous doses, but with a recent relatively low IgG (below 700 BAU). Participants will be tested before and after vaccination with a 4th dose, and followed for 6 months.

As controls, a sub-cohort of similar HCW, who are recruited to the Sheba COVID Cohort study (IRB 8008-20) and are followed monthly with serology tests, and are not receiving the 4th dose. The control group, all of whom signed an informed consent and allowed blood samples to be used for further immunologic studies, will be matched by age, gender, time from 3rd vaccine dose and IgG titers, and will be followed similarly, as by the original 8008-20 protocol.

On recruitment, volunteer will:

1. Receive a detailed explanation and sign the informed consent form (appendix ICF)
2. Fill an initial inclusion/ exclusion criteria questionnaire.
3. Fill a general comorbidity questionnaire (Appendix Q1), additionally they will be screened for COVID-19 symptoms such as fever, cough, anosmia
4. Have up to 40cc blood drawn for all serology and cellular immunity tests.
5. Perform a PCR for SARS-CoV-2 test
6. Receive the 4th dose of mRNA1273 50µg.
7. Will have a physician checkup and followup for 15 minutes after receiving the dose.

Six additional visits will follow as described in the research timeline:

ELIGIBILITY:
Inclusion Criteria:

1. Age: Volunteer must be at least 18 years of age, at the time of signing the informed conset.
2. Sex: Male or Female. All female volunteers of reproductive age will be requested to use contraceptive measures for the two months following enrolment.
3. Received 3 doses of BNT162b2 with the 3rd dose at least 4 months previously.
4. Have a serology test within the previous 3 months of 700 BAU or less.
5. Responded to the previous vaccine doses, i.e. at least one IgG>100.
6. Medical Conditions: Volunteers with any medical condition are allowed, as long as they adhere to the criteria above.
7. Agreed to attend all visits and signed the informed consent - -

Exclusion Criteria:

1. Had previous SARS-CoV-2 infection (detected by either PCR, anti-S IgG before the 1st vaccine dose, anti-N IgG at any stage).
2. Had an allergic response to any of the previous BNT162b2 doses.
3. Has history of myopericarditis.
4. Report that they do not feel well or have a fever on the day of vaccination.
5. Pregnant on day of recruitment -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-01-05 (Actual); Primary Completion 2024-07-04 (Estimated); Study Completion 2024-07-04 (Estimated)

PRIMARY OUTCOMES:
Geometric mean of antibody titers of each arm, on each time point | 6 months
  Serology tests including IgG, neutralization, Tcell activity. These outcomes will be compared between pre- and post- 4th dose, from day 0 to day 180 (6 month), as well as with those outcomes in the control group as well as in Study 8980-21 of participants recieving BNT162b2 as a fourth dose. One blood sample is drawn for all outcome measurments (IgG, neutralization, Tcell activity), which represent the outcome of immunogenecity. IgG is measured in Binding Antibody Units (BAU), minimum value 0, maximum value 50000. Neutralizing antibodies are measured in International units (IU),minimum value 1, maximum value 262144. T cells activity is measured in T cells activity/1 million cells, minimum value 0, maximum value 1000. The higher the score the higher amount of antibodies and t cells activity.
Solicited and unsolicited adverse events | 6 months
  Solicited adverse events will be recorded by questionnaires on days 5,7, 14 and 21. Unsolicited adverse events will be recorded during the whole study period, till day 180 (6 months). Adverse event reporting of vaccinated individuals by an electronic survey that will be filled from visit 2, during each of the first 3 visits.
  Serious adverse events will be defined as any adverse event that resulted in death, hospitalization, permanent damage, required treatment in the emergency room or was life threatening, and will be followed up to 6 months. Higher score reported via the questionnaire represents more serious adverse events.

SECONDARY OUTCOMES:
Commulative incidents of infections in each arm | 6 months
  Rate reduction of infections as well as symptomatic disease in the intervention group, compared to that in the control as well as that in the parallel intervention study with BNT162b2

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Yes
Unidentified data will be available after publication of the results (all IPD that underlie results in a publication)
Supporting Information: Study Protocol, SAP
Time Frame: will be available upon publication of results.
Access Criteria: upon request

REFERENCES:
- [Derived] Canetti M, Barda N, Gilboa M, Indenbaum V, Mandelboim M, Gonen T, Asraf K, Weiss-Ottolenghi Y, Amit S, Doolman R, Mendelson E, Harats D, Freedman LS, Kreiss Y, Lustig Y, Regev-Yochay G. Immunogenicity and efficacy of fourth BNT162b2 and mRNA1273 COVID-19 vaccine doses; three months follow-up. Nat Commun. 2022 Dec 13;13(1):7711. doi: 10.1038/s41467-022-35480-2. PMID 36513665